CLINICAL TRIAL: NCT02021539
Title: The Prognostic Value of Cervical Elastography for Identifying Patients at Risk for Preterm Delivery
Acronym: ElastoMAP
Status: Terminated | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/VL-01
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Obstetric Labor; Labor Onset; Obstetric Labor, Premature
Keywords: Elastography of the cervix; Cervical elastography; Predicting delivery
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Tocolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population consists of pregnant women presenting between the 24th and 34th week of pregnancy, with uterine contractions associated with cervical changes objectified by ultrasound examination of the cervix (5-25mm) who consult for obstetric emergencies (both single or multiple pregnancies can be included).
  Intervention : Cervical ultrasound +elastography 1 Intervention : Vaginal fibronectin measurement Intervention : Tocolytic treatment for 2 hours Intervention : Cervical ultrasound +elastography 2
  Interventions: Procedure: Cervical ultrasound +elastography 1; Biological: Vaginal fibronectin measurement; Drug: Tocolytic treatment for 2 hours; Procedure: Cervical ultrasound +elastography 2

INTERVENTIONS:
Procedure: Cervical ultrasound +elastography 1 — Included patients will have a cervical ultrasound upon arrival in the maternity ward. This latter exam will include elastographic measurements, and will be followed by a vaginal fibronectin measurement. Patients will then be treated via a tocolytic (anti-contraction treatment), and two hours later a second cervial ultrasound including elastographic measures will be performed.
Biological: Vaginal fibronectin measurement — Included patients will have a cervical ultrasound upon arrival in the maternity ward. This latter exam will include elastographic measurements, and will be followed by a vaginal fibronectin measurement. Patients will then be treated via a tocolytic (anti-contraction treatment), and two hours later a second cervial ultrasound including elastographic measures will be performed.
Drug: Tocolytic treatment for 2 hours — Included patients will have a cervical ultrasound upon arrival in the maternity ward. This latter exam will include elastographic measurements, and will be followed by a vaginal fibronectin measurement. Patients will then be treated via a tocolytic (anti-contraction treatment), and two hours later a second cervial ultrasound including elastographic measures will be performed.
Procedure: Cervical ultrasound +elastography 2 — Included patients will have a cervical ultrasound upon arrival in the maternity ward. This latter exam will include elastographic measurements, and will be followed by a vaginal fibronectin measurement. Patients will then be treated via a tocolytic (anti-contraction treatment), and two hours later a second cervial ultrasound including elastographic measures will be performed.

SUMMARY:
The hypothesis tested is that the physical changes associated with cervical ripening result in a detectable decrease in rigidity. The main objective of this study is therefore to determine whether the measured elastographic rigidity of cervical tissues in addition to cervix size can be used to predict delivery within the next 48 hours (creation of a prognostic score).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A-To compare the prognostic qualities of elastography scores and fetal fibronectin measurements for predicting the risk of delivery in the next 48 hours.

B-To evaluate the economic impact of introducing elastographic and fibronectin measures during consultatios for obstetric emergencies from the point of vue of the French social security system and the hospital.

C-To evaluate the prognostic value of elastographic measurements in the subgroup twins.

D-To study elastography variation according to patient outcomes.

E-Evaluate the reproducibility of intra-and inter-rater elastographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Pregnant women presenting between the 24th and 34th week of pregnancy, with uterine contractions associated with cervical changes objectified by ultrasound examination of the cervix (5-25mm)
* Single or multiple pregnancy

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient has lost her water (placental rupture)
* History of cervical surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of pregnant women presenting between the 24th and 34th week of pregnancy, with uterine contractions associated with cervical changes objectified by ultrasound examination of the cervix (5-25mm) who consult for obstetric emergencies (both single or multiple pregnancies can be included).
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Ultrasound measure of the cervix (mm) | Day 0
Ultrasound measure of the cervix (mm) | Day 2
Elastography score | Day 0 or within 12 hours
  The score ranges from 0 to 10.

SECONDARY OUTCOMES:
Elastography score | after 2 hours of tocolytic treatment on day 0
  Score ranges from 0 to 10
Vaginal fetal fibronectin | Day 0
Vaginal fetal fibronectin | Day 2
Avoidable hospital costs | Hospital discharge (expected maximum of 20 days)
Was the first ultrasound/elastography carried out while the patient was already on tocolytics? yes/no | Day 0 or 1

OTHER OUTCOMES:
Patient age | baseline (day 0)
Body mass index | baseline (day 0)
Number of previous vaginal deliveries | baseline (day 0)
Pregnancy term | baseline (day 0)
Prescribed treatment (rest, hospitalization, medications) | baseline (day 0)
Delay between first cervical ultrasound upon patient arrival and first ultrasound with elastography | Day 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France